CLINICAL TRIAL: NCT03753230
Title: Clinical Qualification Study of Electroencephalographic Mobile Equipment for the Capture of Emotions
Acronym: QUAdEMCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: API/2018/92
Record Dates: First submitted 2018-11-20; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Musical Emotions
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EEG Device 1 (Experimental): Participants are listening to music while their neural activity is recorded with Emotiv Epoc+
  Interventions: Device: Electroencephalography
- EEG Device 2 (Experimental): Participants are listening to music while their neural activity is recorded with g.tec
  Interventions: Device: Electroencephalography
- High density EEG (Active Comparator): Participants are listening to music while their neural activity is recorded with high density 256 electrodes EEG Geodesic
  Interventions: Device: Electroencephalography

INTERVENTIONS:
Device: Electroencephalography — Cerebral measurements from electroencephalography devices while music is presented to the participant

SUMMARY:
The study aim to determine the reliability of various EEG wireless headsets. Their signal will be compared to standard high-density EEG recording during music listening.

ELIGIBILITY:
Inclusion Criteria:

* Right handed healthy people
* sensitive to "music chill" (Barcelona Reward music Questionnaire>50)
* having given their participation agreement
* individual with health insurance coverage.

Exclusion Criteria:

* Pregnant women
* individuals in "exclusion period" of another study
* subjects with auditory deficits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Quality and spatial/temporal coherence in oscillatory responses patterns recorded with EEG wireless headsets (Emotiv and g.tec) and with the EEG high density gold standard | Up to 2 weeks
  Brain activity will be recorded continuously during musical extract listening. The coherence of EEG activity between the three different devices on similar electrodes will be measured and compared for several brainwaves (delta, theta, alpha, beta, gamma)